CLINICAL TRIAL: NCT01694238
Title: Circular, Mesh Enforced or Cruciate Incision in the Abdominal Wall Fascia for coloStomy Construction - A Randomised Trial
Brief Title: A Randomized Trial on the Technical Aspects of Stoma Construction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: The Swedish Society of Medicine (Other); The Swedish agreement concerning research and education of doctors (Unknown)
Responsible Party: Principal Investigator, Eva Angenete, M.D., Ph.D., senior consultant surgeon, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Stoma-Const
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Colostomy; Colorectal Neoplasm; Diverticulitis
Keywords: Colostomy; Surgical technique
MeSH Terms: conditions — Colorectal Neoplasms; Diverticulitis

ARMS (3):
- Cruciate incision (Active Comparator): Cruciate incision in the abdominal wall fascia
  Interventions: Procedure: Cruciate incision
- Circular incision (Experimental): Circular incision in the fascia
  Interventions: Procedure: Circular incision
- Mesh enforced cruciate incision (Experimental): Mesh enforcement and then cruciate incision in the abdominal wall fascia
  Interventions: Other: Mesh enforced cruciate incision

INTERVENTIONS:
Procedure: Cruciate incision
  Arms: Cruciate incision
Procedure: Circular incision
  Arms: Circular incision
Other: Mesh enforced cruciate incision
  Arms: Mesh enforced cruciate incision

SUMMARY:
An investigation on the difference in stoma hernia frequency related to surgical technique when incising the fascia. All patients planned for elective colostomy formation are to be included. Patients undergoing rectal resection with a TME and a colostomy (Hartmann's procedure) for rectal cancer, abdominoperineal resection for rectal cancer or diverting colostomy for any reason are all included.

The three groups for randomization are:

A. circular incision in the abdominal wall fascia B. cruciate incision in the abdominal wall fascia C. mesh enforced cruciate incision in the abdominal wall fascia Primary endpoint is the parastomal hernia rate within 12 months from index surgery. Secondary end-points include clinical variables, re-admission and/or re-operation due to any stoma complication, quality of life and health economy analyses, at 12 months.

DETAILED DESCRIPTION:
Colostomy formation has been a standard surgical procedure for more than 100 years. Initially the quality of life for stoma patients was all but good, as the appliances to collect the feces were cumbersome, smelly and did not ensure non-leakage. As late as in the 60-ies bandages were still primitive(1). Gradually these problems have decreased as techniques for bandages have improved. A well functioning colostomy may in itself not negatively affect the patient's Quality of Life (QoL)(2), although thorough information and support from stoma care nurses is of utmost importance (3). However, this can only be said if the stoma is well functioning and if the complications are kept to a minimum. The complication rate after stoma formation is still considerable, with figures of 21-70% (4, 5) and studies have shown that adequate height; type of stoma, BMI, emergency surgery and gender may be of importance in reducing the risk of complications both in the short and long-term (6-8).

The surgical technique of stoma formation is only partly evidence based. There are few studies directed at technical details about stoma construction and their future impact on stoma function, apart from the importance of the stoma height (6). One study has tested to standardize the skin incision to 2/3rds of the width of the bowel (9), although the actual impact of this on the functional outcome of the stoma was not presented.. In the surgical literature a cruciate incision in the fascia and extraction of the bowel through a hole sufficient in size is a short description of the surgical technique (10). In clinical practice sufficient size of the hole has often been equal to "two fingers-width", is commonly used, which refers to the width of the surgeon's fingers, a fairly inexact measurement. A pilot study from Sahlgrenska University Hospital has found that this clinical practice for the most part results in a skin incision diameter of 50% of the bowel width.

There have been discussions regarding the placement of the stoma and effects on hernia incidence, whether in the obliquous muscle or the rectus abdominis (11) or if the bowel should take an extraperitoneal route (ad modum Goligher) or not (12). No studies have been sufficient in design or size to thoroughly answer the question.

Parastomal hernia is a long-term complication that is common, in the literature figures up to almost 50% have been reported (13, 14). Attempts to reduce the rates of parastomal hernias have been made in the last few years with a placement of a mesh, at the construction of the stoma, (15-19). This practice has not been universally accepted, in part due to a hesitance in the surgical society because of the risk of infections with foreign body material, and partly due to that most studies are underpowered for their main outcome variable. Another suggestion for the basic construction of the stoma has been to make a circular incision in the fascia instead of a cruciate, but this has not been documented in any studies. It has been described in conjunction with use of circular stapling devices in the skin, no hernias were found, however the patient numbers were small (20). It is apparent that further studies are most welcome.

The evaluation of parastomal hernias has been discussed. Janes et al. used clinical examination in their studies (16, 17), and confirmed in a later study that the concurrence with a CT-verified parastomal hernia was (21) sufficient if performed in a prone position. Another recent study found that results from a CT-scan was not correlated with patient symptoms (22). Other studies have evaluated the use of ultrasound and found it feasible (23). The conclusion must be that evaluation of parastomal hernias may be difficult and must be standardized in a study.

The hypothesis to be tested in this study is that a circular incision or mesh enforced cruciate incision in the abdominal wall fascia with a diameter of 50% of the width of the patients left colon results carries less risk of parastomal herniation than a cruciate incision where the each of the arms measure 1/2 of the diameter of the patients left colon.

The aim of this trial is to compare the parastomal hernia formation within 12 months after stoma surgery between circular, mesh enforced cruciate and cruciate incision.

ELIGIBILITY:
Inclusion Criteria:

* presenting with a cancer or other conditions for which an elective surgical procedure is planned and includes a permanent colostomy formation
* possible to operate in regard to concomitant disease
* giving informed consent to participate

Exclusion Criteria:

* Not possible to operate due to concomitant disease
* Participation in other randomized trials in conflict with the protocol and end-points of the Stoma-Const trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2013-06; Primary Completion 2017-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Stoma hernia frequency at 12 months | 12 months
  The frequency of stoma hernia at 12 months measured either by clinical examination or CT scan

SECONDARY OUTCOMES:
Readmission | 12 months
  Number of readmissions in the two groups
Postoperative infections | 12 months
  Postoperative infections at 12 months
Total hospital stay | 12 months
  The total number of days in hospital during 12 months
Other complications | 12 months
  The number and type of complications during 12 months postoperatively
30 day mortality | 30 days
  30 day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Eva Angenete, M.D., Ph.D., Principal Investigator — Sahlgrenska University Hospital, Sahlgrenska Academy, Gothenburg University and SSORG - Scandinavian Surgical Outcomes Research Group
Locations (1):
- Sahlgrenska University Hospital/östra, Gothenburg, Sweden

REFERENCES:
- [Derived] Correa Marinez A, Erestam S, Haglind E, Ekelund J, Angeras U, Rosenberg J, Helgstrand F, Angenete E. Stoma-Const--the technical aspects of stoma construction: study protocol for a randomised controlled trial. Trials. 2014 Jun 27;15:254. doi: 10.1186/1745-6215-15-254. PMID 24970570